CLINICAL TRIAL: NCT01735162
Title: Prospective Study of Acute Kidney Injury in Critically Ill Children Predicted by Renal Angina and Urinary Biomarkers
Brief Title: Study of the Prediction of Acute Kidney Injury in Children Using Risk Stratification and Biomarkers
Acronym: AKI-CHERUB
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Rajit Basu, MD, F.A.A.P., Director, Center for Acute Care Nephrology, Children's Hospital Medical Center, Cincinnati
Other Study IDs: CIN001-AKI-CHERUB
Record Dates: First submitted 2012-11-12; First posted 2012-11-28 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Renal Angina; Acute Kidney Injury
Keywords: Renal angina; AKI; Pediatric Intensive Care
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary samples, intended for discard so waiver of consent obtained. Urine samples spun and frozen at -80C. Samples to be run for biomarker ELISA kits.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Very high risk: Very high risk PICU patients are on mechanical ventilation and at least one inotrope or vasopressor at time of admission
- High Risk: High risk PICU patients have a history of transplantation (solid organ or bone marrow)
- Moderate risk: Moderate risk PICU patients are all other admissions to the ICU (may have either mechanical ventilation or inotropy/vasopressor use but not both). Cannot have a history of transplant. Minimum expected stay 48 hours.

SUMMARY:
Acute kidney injury (AKI) is a common clinical event with severe consequences. In the pediatric intensive care unit (PICU), AKI occurs in almost 10% of all patients and evidence suggests that children are dying not just with AKI, but from AKI. Unfortunately, the treatment for AKI is limited to a great extent by delayed diagnosis. Reliance on markers of kidney injury that change only when significant damage has already occurred has rendered potential therapies ineffective. For this reason, identification of new markers of AKI that change early in the course of injury is paramount. While new AKI biomarkers have been identified, their performance in the general PICU population is variable. The investigators recently proposed the concept of 'renal angina' as a way to risk stratify patients in the ICU for AKI risk. In the AKI-CHERUB study, the investigators propose to study renal angina in PICU patients alone and in combination with urinary biomarkers for AKI prediction. The investigators hypothesize that renal angina will increase the predictive precision of urinary biomarkers for AKI.

DETAILED DESCRIPTION:
Reliance on serum creatinine and urine output for diagnosis of acute kidney injury (AKI) has limited the ability of potential therapeutic measures to be effective. The investigators' recent proposition of the renal angina construct aims to improve and expedite AKI diagnosis through use of risk stratification. An apt parallel is the profound outcome change that has been effected in acute coronary syndrome through targeted troponin measurements in patients with both risk factors and clinical symptoms of coronary ischemia. Novel AKI biomarkers will struggle to gain widespread use until their performance in patients of varying degrees of AKI risk can be balanced with their cost and availability. The investigators hypothesize risk stratification using renal angina (ANG) identifies children at-risk vs. not at-risk for AKI, focusing subsequent biomarker measurement to "rule out" AKI only in children with ANG, increasing biomarker predictive precision. This study is significant because it represents the next step in the vertical integration of AKI biomarkers into routine clinical practice to guide their use rationally. The identification of at-risk patients to guide appropriate biomarker use is high-impact because it will make implementation of preventive and supportive therapies for AKI more effective; data from this study would serve to provide the indications to the Food and Drug Administration (FDA) for biomarker use in critically ill children. The study is innovative because it is the first prospective attempt to study the predictive performance of biomarkers AKI in the PICU population using ANG stratification. The investigators will observe all children admitted to the PICU with an expected length of stay > 48 hours. Urine will be collected from these children and levels of neutrophil gelatinase associated lipocalin (NGAL), interleukin-18 (IL-18), liver-fatty acid binding protein (l-FABP), and kidney injury molecule-1 (KIM-1) will be measured. Renal angina will be assessed at time of admission. Primary outcome will be presence of AKI (as measured by Kidney Diseases Improving Global Outcome (KDIGO) Class 2 or greater) at hospital day 3.

ELIGIBILITY:
Inclusion Criteria:

* Minimum stay 48 hours
* Indwelling urinary catheter

Exclusion Criteria:

* History of renal disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All children admitted to a tertiary children's hospital pediatric intensive care unit with an expected length of stay > 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | At day 3 of PICU admission
  Development of AKI by KDIGO Stage 2 criteria (Creatinine > 200% baseline)

SECONDARY OUTCOMES:
PICU length of stay | 60 days
  Observational assessment of duration of length of stay in PICU from time of renal angina assessment

OTHER OUTCOMES:
Mortality | 60 day
  Incidence of death within 60 days of ICU admission
Renal replacement therapy | During ICU stay
  We will use a dichotomization (yes/no) of whether renal replacement therapy was used in each patient until ICU discharge or death, whichever came first, followed up to 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Goldstein, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Goldstein SL. Acute kidney injury biomarkers: renal angina and the need for a renal troponin I. BMC Med. 2011 Dec 21;9:135. doi: 10.1186/1741-7015-9-135. PMID 22189039
- [Background] Basu RK, Chawla LS, Wheeler DS, Goldstein SL. Renal angina: an emerging paradigm to identify children at risk for acute kidney injury. Pediatr Nephrol. 2012 Jul;27(7):1067-78. doi: 10.1007/s00467-011-2024-5. Epub 2011 Oct 20. PMID 22012033
- [Background] Goldstein SL, Chawla LS. Renal angina. Clin J Am Soc Nephrol. 2010 May;5(5):943-9. doi: 10.2215/CJN.07201009. Epub 2010 Mar 18. PMID 20299370
- [Derived] Gist KM, Selewski DT, Brinton J, Menon S, Goldstein SL, Basu RK. Assessment of the Independent and Synergistic Effects of Fluid Overload and Acute Kidney Injury on Outcomes of Critically Ill Children. Pediatr Crit Care Med. 2020 Feb;21(2):170-177. doi: 10.1097/PCC.0000000000002107. PMID 31568240
- See also: Center for Acute Care Nephrology — http://www.cincinnatichildrens.org/service/c/cacn/default/